CLINICAL TRIAL: NCT03184116
Title: Reducing Violence Among High Risk African American Men in Focused Deterrence Program Through Individual Support
Brief Title: Effects of Individual Intervention for Men in Focused Deterrence Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Sylvie Mrug, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Violence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual intervention (Experimental): Individual intervention using cognitive-behavioral principles
  Interventions: Behavioral: Individual intervention
- Control (No Intervention): No additional intervention

INTERVENTIONS:
Behavioral: Individual intervention — Individual intervention based on a cognitive-behavioral program Reasoning & Rehabilitation
  Arms: Individual intervention

SUMMARY:
This project will implement and evaluate a community-based intervention to improve individual outcomes in violence-related injuries and homicide. Young African American men participating in a focused deterrence program (the Birmingham Violence Reduction Initiative, BVRI) will be randomized to receive an additional individual intervention based on the cognitive-behavioral Reasoning and Rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* African American male identified as at high risk for violence by the Birmingham Violence Reduction Initiative

Exclusion Criteria:

* Mental retardation, serious mental illness (eg, psychosis)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Violence | 6 months
  involvement in violent incidents based on police records and self-report

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No